CLINICAL TRIAL: NCT07201974
Title: iWalk in VR: Integration of Virtual Reality-based Locomotor Rehabilitation in Clinical Care
Brief Title: Virtual Reality for Post-Stroke Gait Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Anouk Lamontagne, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-50-2026-2380
Record Dates: First submitted 2025-09-09; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Rehabilitation; Intervention; Community Walking; Virtual Reality; Clinical care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Intervention study involving a single group, multiple-pre, multiple-post, sequential design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR training (Experimental): Participants will engage in a 4-week VR intervention that comprises of 1-hour training sessions, 2 times/week.
  Interventions: Other: Virtual Reality Training

INTERVENTIONS:
Other: Virtual Reality Training — The VR intervention involves the intensive practice of community ambulation skills. The training sessions will be performed in a virtual environment. During the intervention, stroke participants will be invited to practice different dimensions of community ambulation, such as postural transitions, avoiding other pedestrians, dual-task walking, etc.

SUMMARY:
The goal of this clinical trial is to: (1) implement and test the feasibility of a new VR-ODT intervention offered as part of usual therapy time of patients with a sub-acute stoke; (2) explore the acceptability of the intervention from the perspective of clinicians and patients and; (3) implement measures to optimize the uptake and sustainability of the intervention within the clinical setting.

Participants will engage in a personalized VR-ODT training for 4 weeks (2X 1hr/week) targeting six well-established community walking demands related to (1) walking speed and (2) distance; (3) postural transitions; (4) obstacle avoidance; (5) dual-task walking and; (6) a combination of demands 1-5. For each demand, patients will progress through levels of increasing difficulty according to personalized goals and success criteria.

DETAILED DESCRIPTION:
The project involves the VR-ODT set-up and intervention aimed at improving community walking in stroke survivors, to be implemented and tested within the clinical setting. The set-up comprises of a VR headset (HTC Vive) and an ODT (Infinadeck- to our knowledge the only one in Canada) allowing users to walk at self-selected speed in any direction (360 degrees) in a virtual environment representing a shopping mall in Montreal and nearby streets. Stroke individuals with an altered walking capacity (speed: 0.3 - 0.95m/s) will be recruited from the JRH in- and outpatient programs for 12 consecutive months.

Feasibility (Obj. 1) will be examined using the following measures collated post intervention: number of eligible vs. referred patients and treating clinicians involved; patient and clinician characteristics; adherence to the intervention and adverse events. Perceived mental and physical demands (NASA Tax Load Index), sense of presence (Single- Item Presence Questionnaire) and cybersickness (Simulator Sickness Questionnaire) will also be assessed. Acceptability (Obj. 2) patients and clinicians will be assessed using a Technology Acceptance Model Questionnaire that includes questions related to perceived ease of use and usefulness, as well as with open-ended questions. To optimize uptake and sustainability (Obj. 3), two clinicians (1 occupationnel therapist & 1 physiotherapist) from the JRH stroke program will be trained as clinician-champions (CC) on using the VR-ODT intervention and supporting other clinicians with intervention delivery. The CC, in collaboration with the team, will generate instructional materials (written and video) that detail the intervention, targeted users and step-by-step procedures for clinical use. The CC will also be involved in demonstrations (X2) on the use of the intervention for clinicians. They will be the resource for any question or required assistance with the VR-ODT set-up & intervention.

ELIGIBILITY:
Inclusion Criteria:

People with chronic stroke and persistent deficits in walking / visual-perceptual / cognitive capacities. They can be male or female, aged from 40 to 74 years, with normal/corrected visual and auditory acuity, and present with:

* First-ever supratentorial unilateral stroke 9-24 months ago (such chronicity will ensure steady-state mobility without long-term disuse-related changes
* Mild-to-moderate hemiparesis (Chedoke McMaster Stoke Assessment stages 4/7-6/7 on postural control, leg & foot)
* Ability to walk independently with/without walking aids for at least 1 min at 0.3-0.95 m/s (such a speed range indicates mobility not sufficient for functional community ambulation: shopping ~1.1m/s, street crossing ~1.2 m/s)
* Intact or mildly affected cognitive function (Montreal Cognitive Assessment scores ≥ 22/30)
* Intact to moderately affected visual-perceptual function (positive scores on a maximum of 3/6 tasks on the Behavioural Inattention Test)

Exclusion Criteria:

* Subjects with comorbidities interfering with walking
* Subjects with comorbidities interfering with visual perception
* Subjects without medical clearance for exercise

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: adherence to intervention - number of completed sessions | 2x/week over the 4-week intervention
  Training logbook filled by clinicians
Feasibility: presence of adverse or undesirable effects during the intervention | Post-Intervention (week4)
  Assesses by systematically collecting any occurrence of adverse/unwanted events (falls, injuries, fatigue, etc). Collected with open-ended questions.
Feasibility: Number of participants recruited in each program | Pre-intervention (week0)
  Number of early discharged participants vs. outpatient program participants
Feasibility: Characteristics of stroke participants: age | Pre-intervention (week 0)
  Collected via medical charts
Feasibility: Characteristics of stroke participants: sex | Pre-intervention (week 0)
  Collected via medical charts
Feasibility: Characteristics of stroke participants: gender | Pre-intervention (week 0)
  Collected via medical charts
Feasibility: Characteristics of stroke participants: walking capacity | Pre-intervention (week 0)
  Collected via medical charts. According to physiotherapy evaluations, walking capacity is characterized as severely, moderately or mildly affected.
Feasibility: Characteristics of stroke participants: cognitive function | Pre-intervention (week 0)
  Collected via medical charts. According to occupationnal therapy evaluations, cognitive fonction is characterised as severely affected, moderately affected, mildly affected, or intact.
Feasibility: Characteristics of stroke participants: visual-perceptual function | Pre-intervention (week 0)
  Collected via medical charts. According to occupationnal therapy evaluations, visual-perceptual function is characterised as severely affected, moderately affected, mildly affected, or intact.
Feasibility: Characteristics of clinicians | Pre-intervention (week0)
  collected via paper-based questionnaire
Feasibility: Number of eligible vs. referred participants | Post-intervention (week4)
  Assessed using the number of participants referred to the study in comparison to the list of admitted patients in the targeted stroke programs.
Feasibility: Perceived mental and physical demands | Post-Intervention (week4)
  Collected using the NASA Tax Load Index. It assesses work load on five 7-point scales. Increments of high, medium and low estimates for each point result in 21 gradations on the scales.
Feasibility: Sense of presence | Post-Intervention (week4)
  Collected with the Single-Item Presence Questionnaire, a brief measure used to assess a participant's sense of presence in a virtual environment. It consists of one question rated on a 7-point Likert scale, ranging from 1 ("not at all") to 7 ("completely").
Feasibility: Presence of cybersickness | Post-Intervention (week4)
  Collected via the Simulator Sickness Questionnaire, used for assessing symptoms of motion or simulator sickness following exposure to virtual environments. It includes 16 symptoms rated on a 4-point scale from 0 ("none") to 3 ("severe"), covering nausea, oculomotor discomfort, and disorientation.
Acceptability of the intervention | Post-intervention (Week4)
  Assesses using the Technology Acceptance Model based Questionnaire (Tam-Q) based on the technology acceptance model, in which participants (patients and cliniciens) will rate their perception on each dimension using a visual analog scale ranging from 0-56, with higher score representing higher acceptance to the intervention.
Acceptability: Overall experience | Post-Intervention (Week4)
  Investigated through open-ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Anouk Lamontagne, PhD, Principal Investigator — McGill University
Locations (1):
- Jewish Rehabilitation Hospital, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be made available.
Time Frame: Data will be available within 6 months of study completion
Access Criteria: De-identified data will be deposited in a REDCap database and made available to collaborators. Data may also be made available to other researchers via an institutional data repository that will allow adhering to FAIR principles.